CLINICAL TRIAL: NCT00496457
Title: A Double-Blind, Randomized, Multicenter Study With 500 mg QD of TRO19622 Versus Placebo in Patients With Painful Peripheral Diabetic Neuropathy
Brief Title: Efficacy Study With 500 mg QD of TRO19622 vs Placebo in Patients With Painful Peripheral Diabetic Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Ergomed GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WN29860; EudraCT Number: 2006-004545-42; TRO19622 CLEQ 1104-1 (Other: trophos id)
Record Dates: First submitted 2007-06-22; First posted 2007-07-04 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Diabetic Neuropathy
Keywords: Diabetic Neuropathy; Painful Peripheral Diabetic Neuropathy; TRO19622; Trophos
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): TRO19622
  Interventions: Drug: Experimental
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: Experimental — Capsules of TRO19622 (125 mg)- Once a day before noon meal during 6 weeks
  Arms: 1
Drug: Placebo comparator — 4 Capsules of PBO per day before noon meal
  Arms: 2

SUMMARY:
The purpose of this study is to assess the efficacy and safety of TRO19622 administered PO daily for 6 weeks compared to placebo administered PO daily in patients with painful peripheral diabetic neuropathy.

DETAILED DESCRIPTION:
Diabetic peripheral neuropathic pain (DPNP) affects approximately 11% of patients with diabetic peripheral neuropathy (DPN). Diabetic neuropathy as the underlying disease is the most common long-term complication of diabetes mellitus estimated to be experienced by a majority of patients at least in a mild manner.

Many patients with (DPNP) do not respond adequately to any individual treatment option. None of the various treatments used can be considered a cure. As a result, although a variety of drugs are available for the treatment of diabetic neuropathic pain, there is a strong need to develop new drugs with greater efficacy and/or fewer adverse effects.

The primary objective of the study is to compare the effect of TRO19622 versus placebo on the 24h neuropathic pain scores during the last 7 days of the 6-week treatment period.

Secondary objectives are to compare the efficacy on neuropathic pain, impact on emotional functioning, safety profile, pain time course, and response rate of TRO19622 versus placebo. Additionally, the pharmacokinetics of TRO19622 will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Be a male >18 years or a post-menopausal female (>60 years of age and at least 1 year of amenorrhea).
* Have painful diabetic neuropathy of >6 months duration and are either pain treatment naive or have important side effects or inadequate relief from their current pain medication.
* Be on current pain medication (prescribed analgesics), stable for at least 3 months before study entry (± 25% dosage of basic pain medication, top-up rescue medication allowed), or pain treatment naive.
* Have stable diabetes, defined as HbA1c <10%, no changes in medication in the previous 3 months, and no new symptoms associated with diabetes in the previous 3 months.
* Have scored >2 points on the Michigan Neuropathy Screening Instrument (MNSI), part B-physical assessment by health professional.
* Have an ECG without any clinically significant abnormality.

The following inclusion criteria should be ascertained at the baseline visit:

* Have measurable pain perception (previous 24h) on the Likert numerical rating scale with a mean≥4.0 points calculated from at least 4 daily measurements over the 7 days immediately prior to the Baseline Visit.
* Have stopped current pain medication at least 14 days prior to the Baseline Visit (except rescue medication).

Exclusion Criteria:

* Be pregnant female, lactating female, or female of child bearing potential (≤60 years of age).
* Have a documented neuropathy of any cause other than those mentioned in the inclusion criteria which might interfere with the assessment of the severity of pain (eg, including, but not limited to, alcoholic, uremic, B12, TSH, chemotherapy, HIV, post surgical, or post-traumatic neuropathy).
* Have other neurological diseases that may produce weakness, sensory loss, or autonomic symptoms, or laboratory test abnormality.
* Have been on pain treatment with strong opioids, more than 4 different drug regimens in the previous year, or a current combination of more than 2 drugs.
* Have a current medication of lipid lowering agents other than statins.
* Have a body mass index (BMI) >40 kg/m2 (obesity grade III).
* Had any surgery within the previous 2 months.
* Have concurrent serious neurological disease (eg, dementia, multiple sclerosis, or any other disease that would impact the ability of the patient to provide consent for study participation).
* Have a recent history (within the previous 6 months) or current evidence of alcohol or drug abuse.
* Have concurrent unstable disease involving any system (eg, advanced carcinoma, myocardial infarction, clinical or ECG signs of myocardial ischemia, cardiac insufficiency i.e.≥ NYHA functional classification class 2, anginal symptoms, current symptoms of CAD, renal impairment, or any other condition that in the opinion of the Investigator would make the patient unsuitable for study participation).
* Participated in any other investigational drug or therapy study within the previous 3 months.
* Changed or interrupted current well-tolerated medication during the previous 3 months.
* Lack of ability or willingness to give informed consent.
* Be possibly dependent on the Investigator or the Sponsor (eg, including, but not limited to, affiliated employee).
* Have hemostasis disorders or a current treatment of anticoagulants.
* Have non-adequate renal and/or hepatic function as follows:

  * Renal - Blood creatinine >1.5X upper limit of normal (ULN)
  * Hepatic - Liver enzymes (ALT and AST) >2 X ULN
* Have a known history of or current cardiac dysrhythmias and / or a known history of or current cardiovascular disease including myocardial infarction except patients with well controlled hypertension only.
* Are not able to comply with regard to the known contraindications, warnings and precautions, drug-interactions and dosing recommendations of paracetamol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2007-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Effect of TRO19622 versus Placebo on the mean 24h neuropathic pain score on the Likert numerical rating scale. | During the last 7 days of the 6-week treatment period

SECONDARY OUTCOMES:
24h Pain time course | Duration of study (within 11weeks after screening)
Analysis for treatment effects: SF-MPQ, SF-BPI, SF36, POMS, Global Impression of Change (Patient / Investigator) | Within 6 weeks of treatment
Adverse events | During the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Abitbol, MD, Study Chair — Trophos, Parc Scientifique de Luminy - Case 931, Luminy Biotech Enterprises, 13288 Marseille Cedex9 - France; Dan Ziegler, MD, Principal Investigator — German Diabetes Center, German Diabetes Clinic, Leibniz Institute at the Heinrich-Heine University, Auf ´m Hennekamp 65, 40225 Dusseldorf, Germany
Locations (31):
- Croatia (4):
  - Univerity Hospital OSIJEK, Department for Diabetes and Endocrinology, J.Huttlera 4, Osijek
  - Genaral Hospital "Josip Bencevic", Internal Medicine Department-Unit for Diabetes, Andrije Stampara 42, Slavonski Brod
  - General Hospital Varazdin, Internal Medicine Department-Unit for Diabetes, Ivana Mestrovica bb, Varaždin
  - University Hospital "Dubrava", University Department for Internal Medicine, Institut for Diabetes, Endocrinology and Metabolic diseases, Avenija Gojka Suska 6, Zagreb
- Germany (10):
  - Diabetes Zentrum Mergentheim - Theodor-Klotzbücher-Straße 12, Bad Mergentheim
  - Diabetologische Schwerpunktpraxis - Wilhelminenstr. 22, Dinslaken-Bruch
  - Deutsches Diabetes Center, Institut für Klinische Diabetologie, Leibniz-Zentrum an der Heinrich-Heine Universität - Auf'm Hennekamp 65, Düsseldorf
  - Klinikum Region Hannover GmbH - Klinikum Hannover Nordstadt - Diabetes Schwerpunktklinik -Medizinische Klinik - Haltenhoffstr. 41, Hanover
  - Universitätsklinikum Heidelberg - Abteilung Innere Medizin I und klinische Chemie - Im Neuenheimer Feld 410, Heidelberg
  - Pro scientia med - Osterweide 10, Lübeck
  - IKFE GmbH - Institut für klinische Forschung und Entwicklung - Parcusstr. 8, Mainz
  - Diabetes Schwerpunktpraxis - Gesundheitszentrum Potsdam GmbH - Hebbelstr. 1A, Potsdam
  - Diabetes Schwerpunktpraxis - Gesundheitszentrum Potsdam GmbH, Hebbelstr. 1A, Potsdam
  - Sophien- und Hufeland-Klinikum gGmbH - Klinik für Neurologie und Klinische Neurophysiologie - Henry-van-de-Velde-Str. 2, Weimar
- Latvia (5):
  - Daugavpils Regional Hospital - Vasarnicu street 20, Daugavpils
  - Zemgale's Diabetes Centre SIA - Zemgales boulevard 15, Jelgava
  - Doctor's Practice in Endocrinology - Meža prospekts 9, 2nd floor, 41.kabinets, Ogre
  - Clinical Research Centre "Riga" - Katrinas dambis 16, Riga
  - Talsu Hospital - Rugena street 7, Talsi
- Poland (6):
  - NZOZ Specjalistyczny Ośrodek, Internistyczno-Diabetologiczny, ul Zamenhofa 10/20, Bialystok
  - Centrum Neurologii Klinicznej - Ul. Dwernickiego 8, Krakow
  - NZOZ Special-Med. Ul. Weteranów 46, Lublin
  - NZOZ MEDICA, ul. Jutrzenki 4, Lublin
  - NZOZ Beta-Med., Plac Wolności 17, Rzeszów
  - Adamiec Rajmund Gabinet Lekarski, ul. Żelazna 34, Wroclaw
- Serbia (6):
  - Centre of Neurology, Clinical Hospital Centre "Dr Dragisa Misovic", Belgrade
  - Clinic for Neurology and Psychiatry, Clinical Hospital Centre "Zvezdara", Belgrade
  - Institute for Endocrinology, Clinical Centre Serbia, Belgrade
  - Neurology Clinic, Military Medical Academy, Belgrade
  - Neurology Department, Clinical Hospital Zemun, Belgrade
  - Center for Neurology, Clinical Centre "Kragujevac", Kragujevac